CLINICAL TRIAL: NCT01763476
Title: Atherectomy and Drug-Coated Balloon Angioplasty in Treatment of Long Infrapopliteal Lesions
Acronym: ADCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herz-Zentrums Bad Krozingen (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Aljoscha Rastan, M.D., Herz-Zentrums Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADCAT(2)
Record Dates: First submitted 2013-01-03; First posted 2013-01-09 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Artery Disease; Occlusion of Artery
Keywords: long infrapopliteal artery lesions; drug-coated balloon angioplasty; atherectomy
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases | interventions — Atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel-coated balloon angioplasty (Active Comparator): Target lesion to be treated with paclitaxel-coated balloon
  Interventions: Procedure: paclitaxel-coated balloon angioplasty
- Atherectomy + paclitaxel-balloon (Active Comparator): Target lesion to be treated with atherectomy (TurboHawk, ev3) and paclitaxel-coated balloon
  Interventions: Procedure: paclitaxel-coated balloon angioplasty; Procedure: atherectomy

INTERVENTIONS:
Procedure: paclitaxel-coated balloon angioplasty — plain balloon angioplasty followed by paclitaxel-coated balloon angioplasty of the target lesion
Procedure: atherectomy — atherectomy (TurboHawk, ev3) followed by paclitaxel-coated balloon angioplasty of the target lesion
  Arms: Atherectomy + paclitaxel-balloon

SUMMARY:
There is both a poor life expectancy and a poor prognosis of limb salvage in those patience with stenoses or occlusions of the lower limb (TASC Consensus). To date only a small number of these patients could be helped through medication or surgery. In fact within the first year following diagnosis of a critical limb ischemia 25% of patients lose their leg and 90% have to undergo a percutaneous transluminal angioplasty (PTA) or bypass surgery. Using PTA for treatment of long infrapopliteal artery lesions, stenosis reoccurs in 70% to 80% of cases 3 months after index procedure. Even the use of drug-eluting balloons leads only to 1-year primary patency rates up to 30%.

The primary objective of this study is to compare the performance of atherectomy followed by a drug-coated balloon angioplasty over drug-coated balloon angioplasty alone in long de-novo infrapopliteal lesions in a prospective, single-center, randomized clinical trial.

DETAILED DESCRIPTION:
This is a single-centre, prospective, randomized study to be conducted in Bad Krozingen (Germany). A total of 80 subjects will be entered into the study and will be randomized on a 1:1 basis to either drug-coated balloon angioplasty or atherectomy and drug-coated balloon angioplasty for infrapopliteal use in subjects with long de-novo stenosis (≥6cm) and symptomatic peripheral artery disease (Rutherford 3, 4, or 5). IVUS of the target lesion prior and after intervention will be performed in 15 patients of each group during index procedure. All subjects will undergo a repeat angiography at 3 months to assess the primary endpoint of In-Segment Binary Restenosis. Follow-up visits are scheduled at 3, 6, 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 50 and 85 years old
* Female of childbearing potential must have a negative pregnancy test within 10 days prior to index procedure and utilize reliable birth control until completion of the 12-month angiographic evaluation
* Clinical diagnosis of symptomatic critical limb ischemia as defined by Rutherford 3, 4, or 5
* Single treatment of de-novo lesion(s) in the tibioperoneal trunk, anterior and/or posterior tibial and/or peroneal artery with a lesion length ≥6cm;
* One vessel in 1 limb may be treated in the study. Additional non-target lesion(s) in remaining non-target vessel(s) can be treated at the physician´s discretion by means of balloon dilation or stent placement
* The total length of target lesion(s) can be maximum 250 mm
* In total a maximum of 4 drug-coated balloons may be used to fully cover the target lesion
* Target vessel is 2.0 and 3.5 mm in diameter (visual estimate)
* Target lesion stenosis is >70% diameter stenosis (visual estimate)
* Guidewire must be across the target lesion and located intraluminally within the distal outflow vessel before study randomization
* Interventions in TASC A and B lesions to restore adequate blood flow, in the same index procedure are allowed. This intervention must be prior to the treatment of the study lesion(s) and successful
* Willing to comply with the specified follow-up evaluation
* Written informed consent prior to any study procedures.

Exclusion Criteria:

* Significant (>50%) stenoses distal to the target lesion (dorsalis pedis artery, plantar arch) that might require revascularization, or impede runoff;
* Angiographic evidence of thrombus within target vessel
* Thrombolysis within 72 hours prior to the index procedure
* In-Stent restenosis or restenosis of a native artery
* Aneurysm in the femoral artery or popliteal artery
* Concomitant hepatic insufficiency, thrombophlebitis, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy
* Recent myocardial infarction or stroke < 30 days prior to the index procedure
* Life expectancy less than 12 months
* Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound of the target limb
* Known or suspected allergies or contraindications to aspirin, clopidogrel bisulfate (Plavix) and ticlopidine (Ticlid), heparin, or contrast agent
* Any significant medical condition which, in the investigator´s opinion, may interfere with the subject´s optimal participation in the study
* The subject is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
primary patency | 6 months
  Primary patency of the target lesion 6 months after index procedure measured by duplex ultrasound (PVR>2.4) and angiography (core lab analysis).

SECONDARY OUTCOMES:
target lesion revascularisation (TLR) | 6 and 12 months
  Need for target lesion revascularisation from baseline to 6 months after index procedure.

OTHER OUTCOMES:
Change in Rutherford-Becker Class | 6 and 12 months
  Change in Rutherford-Becker Class from Baseline to 6 and 12 months after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Franz-Josef Neumann, M.D., Study Director — Universitaets-Herzzentrum Freiburg-Bad Krozingen
Locations (1):
- Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen, Germany

REFERENCES:
- [Derived] Rastan A, Brodmann M, Bohme T, Macharzina R, Noory E, Beschorner U, Flugel PC, Burgelin K, Neumann FJ, Zeller T. Atherectomy and Drug-Coated Balloon Angioplasty for the Treatment of Long Infrapopliteal Lesions: A Randomized Controlled Trial. Circ Cardiovasc Interv. 2021 Jun;14(6):e010280. doi: 10.1161/CIRCINTERVENTIONS.120.010280. Epub 2021 Jun 7. PMID 34092093